CLINICAL TRIAL: NCT07137000
Title: The Effect of Art Therapy on Pain, Anxiety, Hope and Life Satisfaction in Patients Undergoing Colorectal Cancer Surgery: A Randomized Controlled Trial
Brief Title: The Effect of Art Therapy in Patients Undergoing Colorectal Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Büşra Bozkurt, Principal Investigator, PhD Student, Nurse, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Saglik-1000-367
Record Dates: First submitted 2025-07-10; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Colon Cancer; Rectum Cancer
Keywords: surgical nursing; art therapy; pain; anxiety; hope; life satisfaction
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Pain; Anxiety Disorders; Personal Satisfaction | interventions — Art Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): No application will be made to this group, and an evaluation will be made after routine nursing care.
- İntervention group (Art Teraphy) (Experimental): Five different art therapy methods (bead jewelry making, pencil drawing, painting, mandala, clay figure making) will be applied to the people in this group.
  Interventions: Other: Art therapy

INTERVENTIONS:
Other: Art therapy — Five different art therapy methods (making bead jewelry, pencil drawing, painting, mandala, making clay figures) be used for people in this group.
  Arms: İntervention group (Art Teraphy)

SUMMARY:
With the development of modern techniques, art has become important in the provision of health services and has enabled individuals to better recognise themselves and their surroundings. The World Health Organisation states that art has an important role in improving health, preventing and treating diseases. Art therapy is a therapy method that includes various art branches such as music, painting, sculpture and is especially applied to individuals with oncological diseases. The place of art therapy in solving the negative biopsychosocial problems experienced by these individuals before and after surgery is increasing day by day. Although there are studies on art therapy in the literature, there is no study on art therapy after colorectal cancer surgery. Therefore, in this study, it is aimed to examine the effect of art therapy applied to patients undergoing colorectal surgery on pain, anxiety, hope and life satisfaction. The population of the study will consist of patients who underwent colorectal cancer surgery in Marmara University Pendik Training and Research Hospital General Surgery Service between December 2024 and June 2025, and the sample will consist of 96 patients who meet the research criteria and accept to participate in the study. Patients participating in the study will be divided into two equal groups as intervention and control group. In the preoperative period, the patients in the intervention and control groups will be informed about the study, written and verbal consent will be obtained from the participants who accept the study, and the patients will be asked to answer the Patient Identification Form, Herth Hope Scale and Life Satisfaction Scale. The haemodynamic parameters of the patients in the intervention group will be recorded at 14:00 on the 1st, 2nd and 3rd postoperative days, the art therapy activity they have determined will be applied for 40 minutes and the data will be obtained using the Visual Analogue Scale, State Anxiety Inventory, Herth Hope Scale and Satisfaction with Life Scale. Patients in the control group will receive only routine ward care and data will be collected on the same days and hours as the intervention group. The data obtained will be analysed with appropriate statistical methods using SPSS Windows 22.0 software. As a result of the study, it is thought that there will be an improvement in the pain, anxiety, hope and life satisfaction of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 70,
* Planned colorectal cancer surgery,
* Not receiving neoadjuvant treatment (chemotherapy, radiotherapy),
* No diagnosed psychiatric disorder,
* No history of anxiolytic drug use,
* Patients who volunteered to participate in the study

Exclusion Criteria:

* Communication difficulties,
* Mental deficiency,
* Patients with dysfunction or disease in their upper extremities that may prevent them from performing art therapy practices

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
First evaluation- Pain | Patients' pain will be assessed on postoperative days 1, 2, and 3, and on day 10 of discharge. This study is expected to last a total of 6 months, with data collection on the specified days.
  It is a one-dimensional scale used to numerically express pain intensity. This scale consists of a 10-cm-long ruler with the words "no pain" at one end and "unbearable pain" at the other. A score of 0 cm on the scale indicates no pain, while a score of 10 cm indicates unbearable pain. As the score on the scale increases, the pain intensity increases.
Anxiety level | Patients' anxiety will be assessed on postoperative days 1, 2, and 3, and on day 10 of discharge. This study is expected to last a total of 6 months, with data collection on the specified days.
  The anxiety level of the patients will be determined using the State Anxiety Inventory. The scale consists of a total of 20 items. Each item is rated on a four-point Likert-type scale: (1) not at all, (2) a little, (3) a lot, and (4) completely. The total score obtained ranges from 20 to 80. Higher scores indicate higher anxiety.
Hope Levels | It will be evaluated one day before surgery, on the 3rd day after surgery, and on the 10th day after discharge.
  Patients' hope levels will be assessed using the Herth Hope Scale. The scale consists of 30 items and three subscales. Each item has response options of "Not at all appropriate," "Rarely appropriate," "Sometimes appropriate," and "Always appropriate." The total score for the scale ranges from 0 to 90, with higher scores indicating higher hope.
Life Satisfaction | It will be evaluated one day before surgery, on the 3rd day after surgery, and on the 10th day after discharge.
  Patients' life satisfaction will be assessed using the Life Satisfaction Scale. The scale, consisting of five items addressing life satisfaction, has a Cronbach's alpha of 0.88. The possible score range is 5-25. A low score indicates that the individual has low life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gezginci Akpinar, Assoc. Prof., PhD, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No